CLINICAL TRIAL: NCT07236177
Title: Evaluation of a New Method for Detecting Cancer Pathologies by Measuring the Activity of Different Glycosidases in Plasma in Patients With Localized Cancer - Pilot Study: B-GLUCANCER2
Brief Title: B-GLUCANCER2 : A Pilot Study Evaluating a New Method for Cancer Detection by Measuring the Activity of Different Glycosidase Enzymes in the Plasma of Patients With a Localized Cancer.
Acronym: B-GLUCANCER2
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2025-A01440-49
Record Dates: First submitted 2025-09-19; First posted 2025-11-19 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Breast Cancer; Pancreatic Cancer; Pulmonary Cancer; Volatile Organic Compound; Glycosidase Activity; Probes; Tumor Markers, Biological
Keywords: breast cancer; pancreatic cancer; pulmonary cancer; volatile organic compounds; glycosidase activity; localized cancer
MeSH Terms: conditions — Breast Neoplasms; Pancreatic Neoplasms; Lung Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- breast cancer (Active Comparator)
  Interventions: Biological: blood plasma sample
- pancreatic cancer (Active Comparator)
  Interventions: Biological: blood plasma sample
- pulmonary cancer (Active Comparator)
  Interventions: Biological: blood plasma sample
- no cancer (Other): no history of cancer
  Interventions: Biological: blood sampling

INTERVENTIONS:
Biological: blood plasma sample — For each patient, 5ml blood sample will be needed before the surgery and another 5ml blood sample one month after the surgery.
  Arms: breast cancer; pancreatic cancer; pulmonary cancer
Biological: blood sampling — 5ml blood sample for control arm
  Arms: no cancer

SUMMARY:
The goal of this clinical trial is to develop a new cancer diagnostic and prognostic tool based on the dynamic and non-invasive detection of an exogenous volatile molecule, i.e., ethanol, from patients' samples.

Patients' blood plasma will be analyzed with a mixture of volatile organic compound-based probes, each targeting a specific glycosidase. The presence of a given glycosidase in a blood sample would thus be revealed by the detection of an ethanol isotope in the gas phase.

3 groups of patients with localized cancer (breast, prostate, pancreas) will be enrolled, as well as 1 group of patient without any cancer (control group).

For the patients, two 5ml plasma samples will be collected, one before and one after surgery for localized cancers. For healthy volunteers, only one 5ml plasma sample will be collected.

The primary objective will be to compare the levels of glycosidases measured in the blood of patients followed for localized cancer and referred for first surgery compared to control patients without cancer.

ELIGIBILITY:
Inclusion Criteria:

* Group 1: 40 patients with definitively diagnosed, untreated, localized solid breast cancer referred for initial surgical treatment.

Group 2: 40 patients with definitively diagnosed, untreated, localized solid lung cancer referred for initial surgical treatment.

Group 3: 40 patients with definitively diagnosed, untreated, localized solid pancreatic cancer referred for initial surgical treatment.

Group 4: 100 control patients with no cancer diagnosis or history of solid or hematological cancer.

Exclusion Criteria:

* Refusal to participate in the research.
* Patients benefiting from enhanced protection, namely: minors, pregnant/breastfeeding women, persons deprived of their liberty by a judicial or administrative decision, persons staying in a social care facility, adults under legal protection

Specific criteria for groups 1, 2, and 3:

* Cancer patients undergoing oncological treatment.
* Cancer not proven by anatomopathological examination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 220 (Estimated)
Dates: Start 2026-02-03 (Actual); Primary Completion 2028-02-03 (Estimated); Study Completion 2028-03-03 (Estimated)

PRIMARY OUTCOMES:
To compare the levels of glycosidases measured in the blood samples of patients treated for a localized cancer (breast, lung or pancreatic cancer) compared to control patients without cancer. | before surgery and one month after surgery

SECONDARY OUTCOMES:
Compare the seven glycosidase levels in patients with localized breast cancer versus cancer-free control patients. | one month
Compare the seven glycosidase levels in patients with localized pancreatic cancer versus cancer-free control patients. | one month
Compare the seven glycosidase levels in patients with localized lung cancer versus cancer-free control patients. | one month
Compare the seven glycosidase levels according to cancer location (lung versus breast, pancreas versus breast, lung versus pancreas). | one month
Compare glycosidase levels in cancer patients before and after surgery (regardless of location: breast, lung, or pancreatic cancer). | one month

CONTACTS AND LOCATIONS:
Locations (1):
- C.H.U. Poitiers, Poitiers, France

IPD SHARING:
Plan to Share IPD: Yes